CLINICAL TRIAL: NCT03501615
Title: An Early Access Programme for Moxetumomab Pasudotox in Relapsed/Refractory Hairy Cell Leukemia
Acronym: MOXE
Status: Approved for marketing | Type: Expanded Access
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D3143R00002
Record Dates: First submitted 2018-04-10; First posted 2018-04-18 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Relapsed/Refractory Hairy Cell Leukemia
Keywords: Early Access; Leukemia; Hairy cell; Moxetumomab Pasudotox; PNA; Purine analog; BRAF Inhibitor; Rituximab; Pseudomonas-immunotoxin naïve
MeSH Terms: conditions — Leukemia, Hairy Cell; Leukemia | interventions — immunotoxin HA22; HA 22

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Moxetumomab Pasudotox — A recombinant conjugated immunotoxin composed of a disulfide-stabilized anti-CD22 Ig Fv genetically fused to a truncated form of Pseudomonas exotoxin, PE38
  Other Names: CAT-8015, HA22

SUMMARY:
Early Access Programme to provide treatment access to moxetumomab pasudotox for eligible patients with relapsed/refractory hairy cell leukemia

DETAILED DESCRIPTION:
Multicentre Early Access Programme, designed to provide treatment access to moxetumomab pasudotox for eligible patients with relapsed/refractory hairy cell leukemia who are at least 18 years of age, have adequate organ function and are Pseudomonas-immunotoxin naïve. Patients will be administered moxetumomab pasudotox on Days 1, 3 and 5 of each 28-day cycle until documentation of CR or for up to 6 cycles, progressive disease (PD), initiation of alternate therapy or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed HCL or HCL variant with a need for therapy based on at least one of the following criteria:

   a neutrophils < 1.0x 109/L b platelets < 100 x 109/L c hemoglobin < 10 g/dL d symptomatic splenomegaly
2. Pseudomonas-immunotoxin naïve
3. At least 2 prior systemic therapies, including 2 courses of a PNA, or 1 course of either rituximab or BRAF inhibitor following a single prior course of PNA.
4. Age ≥ 18 years.
5. ECOG performance status ≤ 2
6. Adequate organ function as defined below:

   1. total bilirubin ≤ 1.5 mg/dL, unless consistent with Gilbert's (ratio between total and direct bilirubin > 5)
   2. AST and ALT ≤ 3x upper limit of normal (ULN)
   3. alkaline phosphatase < 2.5 ULN
   4. serum creatinine ≤ 1.5 mg/dL or creatinine clearance ≥ 60 mL/min as estimated by the Cockcroft-Gault equation
7. Prothrombin time (PT)/international normalized ratio (INR) or partial thromboplastin time (PTT) < 2.5 ULN, fibrinogen ≥ 0.5 lower limit of normal; if on warfarin, INR < 3.5, if on any other anticoagulation, PT < 2.5 x baseline
8. Ability to understand and the willingness to sign a written informed consent document.
9. Life expectancy ≥ 6 months.
10. Females of childbearing potential who are sexually active with a nonsterilized male partner must use a highly effective method of contraception prior to study entry and for the duration of study participation, and must agree to continue using such precautions for 4 months after completion of moxetumomab pasudotox administration; cessation of contraception after this point should be discussed with a responsible physician. Periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of contraception.

Exclusion Criteria:

1. Have had chemotherapy, immunotherapy or radiotherapy within 4 weeks prior to initiation of treatment. 2. Receiving any other investigational agents. 3. Known brain metastases 4. Retinal or choroidal detachment identified during the screening ophthalmologic evaluation. 5. Pregnant or breastfeeding females. . 6. Positive for Hepatitis B core antibody or surface antigen unless the patient is on Lamivudine or Entecavir and Hepatitis B Viral deoxyribonucleic acid (DNA) load is < 2000 IU/mL. 7. Active second malignancy requiring treatment other than minor resection of indolent cancers like basal cell and squamous skin cancers. 8. Uncontrolled intercurrent illness including but not limited to ongoing or active infection, Symptomatic congestive heart failure, unstable angina pectoris, uncontrolled hypertension, cardiac arrhythmia, malaria infection, or psychiatric illness/social situations that would limit compliance with study requirements. 9. Known human immunodeficiency virus (HIV)-positive patients unless taking appropriate anti-HIV medications with a CD4 count of > 200. 10.History of allogeneic bone marrow transplant. 11.History of both thromboembolism and known congenital hypercoagulable conditions. 12.Uncontrolled pulmonary infection, pulmonary edema 13.Oxygen saturation at rest < 88% measured by pulse oximetry or PaO2

* 55 mm Hg 14.Serum albumin < 2 g/dL 15.Radioimmunotherapy within 2 years prior to enrollment in the study. 16.Absolute neutrophil count (ANC) < 1.0 x 109/L, or platelet count < 50 x 109/L, unless judged by the investigator to be due to underlying disease A patient will not be excluded because of pancytopenia ≥ Grade 3, or erythropoietin dependence, if due to disease, based on the results of bone marrow studies. 17.Patients with < 50% of predicted forced expiratory volume or < 50% of predicted diffusing capacity for carbon monoxide, corrected for hemoglobin concentration and alveolar volume 18.History of thrombotic microangiopathy or thrombotic microangiopathy / HUS. 19.Corrected QT interval (Frederica) elevation > 500 msec (manually over-read by medically qualified person) based on at least two separate 12-lead ECGs. 20.High dose estrogen (defined as > 0.625 mg/day of an estrogen compound). 21.Clinical evidence of disseminated intravascular coagulation (Grade 3- 4).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Nai Shun (Nancy) Yao, MD, Study Chair — MedImmune LLC